CLINICAL TRIAL: NCT00509236
Title: A Multicenter, Randomized Double-Blind Study to Evaluate the Efficacy and Safety of Sitagliptin Versus Glipizide in Participants With Type 2 Diabetes Mellitus and End-Stage Renal Disease Who Are on Dialysis and Who Have Inadequate Glycemic Control
Brief Title: Sitagliptin Versus Glipizide in Participants With Type 2 Diabetes Mellitus and End-Stage Renal Disease (MK-0431-073 AM1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-073; 2007_550 (Other: Merck Study Number)
Record Dates: First submitted 2007-07-27; First posted 2007-07-31 (Estimated); Results first posted 2012-05-03 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus, Type 2; End-Stage Kidney Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Kidney Failure, Chronic | interventions — Sitagliptin Phosphate; Glipizide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin 25 mg (Experimental)
  Interventions: Drug: Sitagliptin
- Glipizide 2.5 mg - 20 mg (Active Comparator)
  Interventions: Drug: Glipizide

INTERVENTIONS:
Drug: Sitagliptin — 25 mg (one 25-mg tablet) once daily
  Other Names: MK-0431
  Arms: Sitagliptin 25 mg
Drug: Glipizide — 2.5 mg (1/2 of a 5-mg tablet) once daily, up to 10 mg twice daily (four 5-mg tablets), for a maximum of 20 mg
  Other Names: Glucotrol
  Arms: Glipizide 2.5 mg - 20 mg

SUMMARY:
The purpose of the study is to compare sitagliptin and glipizide in lowering blood sugar in participants with type-2 diabetes mellitus (T2DM) and end-stage renal disease on dialysis who do not have adequate glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Participant has T2DM.
* Participant is on dialysis on day of signing informed consent.
* Participant is unlikely to conceive or uses acceptable methods of birth control: hormonal contraceptive, intrauterine device (IUD), diaphragm with spermicide, contraceptive sponge, condom, or vasectomy.
* Participant has hemoglobin A1c ≥7% and ≤9% measured at or within 2 weeks prior to Visit 4/Week -2.
* Participant is ≥85% compliant with study medication during the single-blind placebo run-in (as determined by tablet/capsule count) and compliant with diet, exercise and other run-in treatments during the run-in period.

Exclusion Criteria:

* Participant has a history of type 1 diabetes mellitus or a history of ketoacidosis.
* Participant is losing weight in a weight loss program and is not in the maintenance phase (defined as <2 kg weight loss in 2 months), or intends to be involved in weight loss intervention outside that prescribed by the study.
* Participant has a clinically significant hematological disorder (e.g., aplastic anemia, myeloproliferative or myelodysplastic syndromes, thrombocytopenia).
* Participant has cirrhosis or active liver disease.
* Participant has been on dialysis for < 6 months.
* Participant has been diagnosed with a significant cardiovascular disorder and has new or worsening signs or symptoms of congestive heart failure within 3 months of signing informed consent.
* Participant has severe active peripheral vascular disease.
* Participant has a history of malignancy ≤ 5 years prior to signing informed consent, or > 5 years without documentation of remission/cure.
* Participant is under treatment for hyperthyroidism.
* Participant has a hypersensitivity or contraindication to glipizide.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2007-10-19 (Actual); Primary Completion 2011-03-14 (Actual); Study Completion 2011-03-14 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Arjona Ferreira JC, Corry D, Mogensen CE, Sloan L, Xu L, Golm GT, Gonzalez EJ, Davies MJ, Kaufman KD, Goldstein BJ. Efficacy and safety of sitagliptin in patients with type 2 diabetes and ESRD receiving dialysis: a 54-week randomized trial. Am J Kidney Dis. 2013 Apr;61(4):579-87. doi: 10.1053/j.ajkd.2012.11.043. Epub 2013 Jan 24. PMID 23352379

RESULTS

PARTICIPANT FLOW:
Groups:
- Sitagliptin 25 mg: One 25 mg tablet once daily for 54 weeks
- Glipizide 2.5 mg - 20 mg: Between 2.5 mg - 20 mg daily for 54 weeks
Period: Overall Study
Arm/Group | Sitagliptin 25 mg | Glipizide 2.5 mg - 20 mg
Started | 64 | 65
Completed | 47 | 45
Not Completed | 17 | 20
Not completed — Adverse Event | 7 | 9
Not completed — Withdrawal by Subject | 5 | 10
Not completed — Protocol Violation | 3 | 0
Not completed — Excluded Medication | 1 | 1
Not completed — Scheduled Kidney Transplant | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin 25 mg | Glipizide 2.5 mg - 20 mg | Total
Number analyzed (Participants) | 64 | 65 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (9.1) | 58.5 (9.9) | 59.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 28 | 52
  Male | 40 | 37 | 77

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c After Sitagliptin Treatment
Description: Change from baseline in mean hemoglobin A1c after treatment with sitagliptin for 54 weeks. Hemoglobin A1c is the percent of hemoglobin that is glycated. Results for the glipizide arm are not reported in this table because the primary outcome measure is for the sitagliptin arm only.
Time Frame: Baseline / Week 54
Population: Randomized participants. Numbers analyzed excluded participants with either no baseline or no post-baseline measurements. The last observation carried forward (LOCF) method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: Percent hemoglobin A1c
Groups:
- Sitagliptin 25 mg: Participants received one 25 mg tablet once daily for 54 weeks
Arm/Group | Sitagliptin 25 mg
Number analyzed (Participants) | 62
Percent hemoglobin A1c
  Baseline | 7.89 (0.74)
  Week 54 | 7.15 (0.98)
  Change from Baseline at Week 54 | -0.74 (0.95)
Statistical Analysis 1: Comparison: Sitagliptin 25 mg; Model terms: treatment, prior diabetes pharmacotherapy (not on oral antihyperglycemic agent, or on oral antihyperglycemic agent), and a covariate for baseline A1c; Test type: Superiority or Other; p < 0.001, ANCOVA

2. Secondary Outcome: Number of Participants With Symptomatic Hypoglycemic Adverse Events
Description: A symptomatic hypoglycemic adverse event is an episode with clinical symptoms attributed to hypoglycemia, without regard to fingerstick glucose level.
Time Frame: 54 Week Treatment Period + 28 days
Population: All randomized participants.
Measure: Number; unit: Participants
Groups:
- Glipizide 2.5 mg - 20 mg: Participants received between 2.5 mg - 20 mg daily for 54 weeks
Arm/Group | Sitagliptin 25 mg | Glipizide 2.5 mg - 20 mg
Number analyzed (Participants) | 64 | 65
Participants | 4 | 7
Statistical Analysis 1: Comparison: Sitagliptin 25 mg vs Glipizide 2.5 mg - 20 mg; Test type: Superiority or Other; p = 0.336, Miettinen & Nurminen — Miettinen & Nurminen method stratified by prior diabetes pharmacotherapy (not on oral antihyperglycemic agent, or on oral antihyperglycemic agent); Difference in % Affected = -4.8, 95% CI 2-sided [-15.7 to 5.6]

3. Primary Outcome: Number of Participants With Clinical Adverse Events
Description: Reported experiences assessed by investigators as adverse events, excluding data after initiation of glycemic rescue therapy.
Time Frame: 54 Week Treatment Period + 28 days
Population: All randomized participants.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin 25 mg | Glipizide 2.5 mg - 20 mg
Number analyzed (Participants) | 64 | 65
Participants | 53 | 52
Statistical Analysis 1: Comparison: Sitagliptin 25 mg vs Glipizide 2.5 mg - 20 mg; Test type: Superiority or Other; Difference in % Affected = 2.8, 95% CI 2-sided [-10.9 to 16.5]

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Change from baseline in mean Fasting Plasma Glucose after treatment with sitagliptin versus glipizide for 54 weeks.
Time Frame: Baseline / Week 54
Population: Randomized participants. Numbers analyzed excluded participants with no baseline or no post-baseline measurements. The last observation carried forward (LOCF) method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sitagliptin 25 mg | Glipizide 2.5 mg - 20 mg
Number analyzed (Participants) | 60 | 59
mg/dL
  Baseline | 160.3 (48.5) | 167.0 (56.2)
  Week 54 | 135.8 (40.4) | 134.0 (58.2)
  Change from Baseline to Week 54 | -24.5 (47.5) | -33.0 (55.9)
Statistical Analysis 1: Comparison: Sitagliptin 25 mg; Model terms: treatment, prior diabetes pharmacotherapy (not on oral antihyperglycemic agent, or on oral antihyperglycemic agent), and a covariate for baseline FPG; Test type: Superiority or Other; p < 0.001, ANCOVA; Change from Baseline in LS Mean = -26.6, 95% CI 2-sided [-38.0 to -15.3]
Statistical Analysis 2: Comparison: Glipizide 2.5 mg - 20 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Change from Baseline in LS Mean = -31.2, 95% CI 2-sided [-42.6 to -19.9]
Statistical Analysis 3: Comparison: Sitagliptin 25 mg vs Glipizide 2.5 mg - 20 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Difference in LS Means = 4.6, 95% CI 2-sided [-11.5 to 20.7]

5. Secondary Outcome: Change From Baseline in Hemoglobin A1c for Sitagliptin Versus Glipizide Treatment
Description: Change from baseline in least square means hemoglobin A1c after treatment with sitagliptin versus glipizide for 54 weeks. Hemoglobin A1c is the percent of hemoglobin that is glycated.
Time Frame: Baseline / Week 54
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent hemoglobin A1c
Arm/Group | Sitagliptin 25 mg | Glipizide 2.5 mg - 20 mg
Number analyzed (Participants) | 62 | 59
Percent hemoglobin A1c | -0.72 [-0.95 to -0.48] | -0.87 [-1.11 to -0.63]
Statistical Analysis 1: Comparison: Sitagliptin 25 mg vs Glipizide 2.5 mg - 20 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANCOVA; Difference in LS Means = 0.15, 95% CI 2-sided [-0.18 to 0.49]

ADVERSE EVENTS:
Arm/Group | Sitagliptin 25 mg | Glipizide 2.5 mg - 20 mg
Serious Adverse Events (participants affected / at risk) | 23/64 | 22/65
Other Adverse Events (participants affected / at risk) | 33/64 | 37/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin 25 mg (N=64) | Glipizide 2.5 mg - 20 mg (N=65)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 2 (3)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular dysfunstion (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Device malfunction (General disorders) | 2 (2) | 0 (0)
Device occlusion (General disorders) | 1 (1) | 1 (1)
Medical device complication (General disorders) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Arteriovenous fistula site infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 4 (4)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 2 (2)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (3)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (3) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1)
Diabetic foot (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (2) | 2 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 1 (2)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin 25 mg (N=64) | Glipizide 2.5 mg - 20 mg (N=65)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 5 (6)
Vomiting (Gastrointestinal disorders) | 4 (6) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 7 (8)
Urinary tract infection (Infections and infestations) | 5 (6) | 1 (1)
Blood glucose decreased (Investigations) | 11 (37) | 18 (94)
Blood glucose increased (Investigations) | 4 (11) | 5 (13)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (7) | 7 (16)
Headache (Nervous system disorders) | 4 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (7)
Hypertension (Vascular disorders) | 5 (7) | 6 (6)
Hypotension (Vascular disorders) | 4 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Subsequent to the multicenter publication, or 24 months after completion of the study, whichever comes first, an investigator and/or colleagues may publish the results for their study site independently. The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.